CLINICAL TRIAL: NCT03723252
Title: Efficacy and Safety of Dapagliflozin in Non-alcoholic Steatohepatitis: a Multicentre, Randomized, Placebo-controlled Trial
Brief Title: Dapagliflozin Efficacy and Action in NASH
Acronym: DEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Huijie Zhang, Clinical Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2018-127
Record Dates: First submitted 2018-10-23; First posted 2018-10-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Nonalcoholic Steatohepatitis; SGLT-2 inhibitor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin group (Experimental): Participants will receive dapagliflozin 10mg po qd.
  Interventions: Drug: Dapagliflozin
- Placebo group (Placebo Comparator): Participants will receive placebo po qd.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Participants will receive dapagliflozin 10mg po qd
  Arms: Dapagliflozin group
Drug: Placebo — Participants will receive placebo po qd
  Arms: Placebo group

SUMMARY:
This is a multicentre, randomized, placebo-controlled trial to assess the efficacy and safety of dapagliflozin on improving non-alcoholic steatohepatitis as determined by liver biopsies and metabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged≥18 years;
* Non-alcoholic steatohepatitis as determined by liver biopsies within 6 months;
* Patients with T2DM at screening had to have stable glycaemic control (HbA1c <9.5%) .

Exclusion Criteria:

1. Significant alcohol consumption in the past six months (Consumed more than 20 g/day for women or 30 g/day for men);
2. A history of alcoholic liver disease, chronic viral hepatitis, drug-induced hepatitis, autoimmune hepatitis, cirrhosis, and liver cancer;
3. Obstructive biliary disease;
4. Having any medical condition that would affect metabolism (i.e. Cushing syndrome, known hyperthyroidism or hypothyroidism);
5. Poor glucose control (defined as HbA1C≤ 9.5% within 3 months) if diagnosed with T2DM, or taking any antidiabetic medication that would affect metabolism or weight loss (i.e. TZD, GLP-1, DPP-4i or initially using insulin in the past 3 months);
6. Taking any medication (i.e. cortisol, methotrexate)that would affect steatohepatitis for more than two weeks in the past year;
7. Chronic kidney disease or severe impaired renal function (serum creatinine≥ 2.0mg/dl);
8. Serum alanine aminotransferase (ALT) greater than 300U/L
9. A history of Type 1 diabetes;
10. A history of bladder cancer;
11. Women who are pregnant or plan to become pregnant;
12. Serious medical disease with likely life expectancy less than 5 years;
13. Patients who cannot be followed for 24 months (due to a health situation or migration);
14. Participation in other clinical trial in the 30 days before randomization;
15. Patients who are unwilling or unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-28 (Actual)

PRIMARY OUTCOMES:
Improvement in scored liver histological improvement over 12 months | Baseline to 12 months

SECONDARY OUTCOMES:
Resolution of NASH | Baseline to 12 months
  defined as a hepatocellular ballooning score of 0, and lobular inflammation score of 0 or 1) without worsening of fibrosis
Improvement of fibrosis | Baseline to 12 months
  defined as reduction in fibrosis of at least 1 stage) without worsening of NASH
Change in fibrosis score | Baseline to 12 months
Change in each component score in the NAS | Baseline to 12 months
Change in body weight | Baseline to 12 months
Change in waist circumference | Baseline to 12 months
Change in visceral fat | Baseline to 12 months
Change in liver fat | Baseline to 12 months
Change in HbA1C | Baseline to 12 months
Change in blood pressure | Baseline to 12 months
Change in serum lipids | Baseline to 12 months
Change in insulin resistance | Baseline to 12 months
Change in inflammatory markers of NASH | Baseline to 12 months
Change in health related quality of life scores (SF-36) | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Huijie Zhang, MD.PhD., Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin J, Huang Y, Xu B, Gu X, Huang J, Sun J, Jia L, He J, Huang C, Wei X, Chen J, Chen X, Zhou J, Wu L, Zhang P, Zhu Y, Xia H, Wen G, Liu Y, Liu S, Zeng Y, Zhou L, Jia H, He H, Xue Y, Wu F, Zhang H. Effect of dapagliflozin on metabolic dysfunction-associated steatohepatitis: multicentre, double blind, randomised, placebo controlled trial. BMJ. 2025 Jun 4;389:e083735. doi: 10.1136/bmj-2024-083735. PMID 40467095